CLINICAL TRIAL: NCT05693558
Title: A Proof-of-concept Study With NVD-003, an Autologous Osteogenic Bone Graft, in the Treatment of Congenital Pseudarthrosis of the Tibia in Pediatric Patients.
Brief Title: NVD-003 in the Treatment of Congenital Pseudarthrosis of the Tibia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novadip Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVD003-CLN02 CPT; 2022-001282-12 (EudraCT Number)
Record Dates: First submitted 2022-10-26; First posted 2023-01-23 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Congenital Pseudarthrosis of Tibia
Keywords: Tissue Engineered Therapy; bone graft; autologous; pediatric; congenital; non-union; pseudarthrosis; Cellular therapy
MeSH Terms: conditions — Pseudarthrosis

STUDY DESIGN:
Intervention Model Description: A single arm, multi-country, multi-center study in pediatric patients, suffering from congenital pseudarthrosis of the tibia (CPT), treated during the primary surgical intervention with NVD-003, an autologous 3D scaffold free osteogenic graft.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NVD-003 bone graft implant (Experimental): The study includes 2 important surgical procedures, the Adipose Tissue Collection (ATC) and the Grafting Surgery (GS) and 3 stages
  * Stage 1: A screening, adipose tissue collection & NVD 003 manufacturing period.
  * Stage 2: Grafting surgery and 12-month post-GS follow-up period.
  * Stage 3: long-term safety follow-up period (from post-month 12 to month 24).
  Interventions: Biological: NVD-003, an autologous 3D scaffold free osteogenic graft

INTERVENTIONS:
Biological: NVD-003, an autologous 3D scaffold free osteogenic graft — Bone correction and grafting surgery

SUMMARY:
A single arm, multi-country, multi-center study in pediatric patients, suffering from congenital pseudarthrosis of the tibia (CPT), treated during the primary surgical intervention with NVD-003, an autologous 3D scaffold free osteogenic graft.

DETAILED DESCRIPTION:
Congenital pseudarthrosis is a rare disorder of unknown aetiology and variable history that manifests itself as a non-union or pseudarthrosis of fractures that develop spontaneously or following minor trauma. It can be defined as a disorder of the diaphysis which is revealed by either pseudarthrosis at birth or by a pathological fracture presenting in bone with modifications such as bowing, narrowing of the medullary canal or a cyst. Although uncommon, CPT is the most frequently observed type of congenital pseudarthrosis. Its incidence is reported to be between 1:140,000 to 1:250,000 live births.

Autologous bone grafting is considered the gold standard approach as this material vascularizes and integrates with surrounding bone, minimizing the risk of infection, dislodgement, or break-down.

NVD-003 is a scaffold free 3D osteogenic graft derived from autologous adipose stem cells which become embedded in their extracellular matrix and combined with hydroxyapatite/beta-tricalcium phosphate (HA/βTCP) particles.

NVD-003 is intended to promote bone formation, supporting the physiological bone healing process in severe pathophysiological conditions such as hypoxia, lack of mineralized callus formation, bone resorption and low osteogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital pseudarthrosis of the tibia (with or without NF1) and presenting with a non-healing Paley type 3 or 4 fracture.
* Minimum weight of 5kg/11lbs.
* Maximum 2 previous failed surgical orthopaedic interventions to treat the primary CPT fracture.
* Acceptable serology and molecular test results excluding the presence of viruses
* Satisfactory general health condition to undergo surgeries (ATC and GS) with anaesthesia as per local standards.
* The patient's parent(s) and/or legal guardian(s) provided written informed consent and accepted the participation of the patient in the trial.

Exclusion Criteria:

* Bilateral CPT.
* Presence of CPT without a fracture of the tibia (Paley type 1 and 2).
* More than 2 failed surgical attempt(s) to treat the primary tibial fracture.
* Evidence of plexiform neurofibroma of any size or nodular fibroma ≥ 1.2in/3cm on the ipsilateral leg.
* Clinically significant infection at the target grafting site or systemic infection.
* Presence of clinically significant hematologic, renal, hepatic, and coagulation laboratory abnormalities (i.e., CBC, PT/INR, Chem-7, and LFTs, etc.).
* Presence of any auto-immune disease, with exception of well controlled diabetes type 1 or auto-immune thyroid disorders.
* Any history of experimental therapy with another investigational drug within 60 days prior to screening.
* Presence of active tumour.
* Documented metabolic bone disease or any disorder, such as but not limited to osteogenesis imperfecta and osteomalacia, that could interfere with the bone healing and bone metabolism.
* Chronic, ongoing, or planned use of medications that might affect bone metabolism or bone quality such as bisphosphonates, steroids, methotrexate, anticoagulant therapies, immunosuppressant therapy or immunotherapy.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Primary objective: safety short (≤3 months) and mid long-term (>3-12 months): : Descriptive analysis | Up to 12 months post-grafting surgery
  Assess number of patients with NVD-003 related (S)AEs

SECONDARY OUTCOMES:
Long term Safety long-term (>12-24 months): Descriptive analysis | 12-24 months post grafting surgery
  Assess number of patients with NVD-003 related SAEs
Tibial length evaluation | 3-, 6-, 12- and 24-months post-GS
  Assess evolution tibial length (using CT-Scan)
Bone formation | 3-, 6-, 12- and 24-months post-GS
  Assess changes in bone formation (Using Lane and Sandhu Scoring on CT-Scan)
Bone remodeling | 3-, 6-, 12- and 24-months post-GS
  Assess changes in bone remodeling (using Lane and Sandhu Scoring on CT-scan)
  Based on Dual Energy CT-scan (DECT or Spectral CT), information of low- and high-energy photons is collected, allowing to uncover differences in energy-dependent attenuation, facilitating composition of NVD 003 and surrounding tissue and define bone mineral density) at 3-, 6-, and 12-months post-GS
Bone union | 3-, 6-, 12- and 24-months post-GS
  Assess changes in bone union (using Lane and Sandhu Scoring on CT-scan)

CONTACTS AND LOCATIONS:
Overall Officials: Philip McClure, MD, Principal Investigator — International Center for Limb Lengthening Baltimore; Pierre-Louis Docquier, Principal Investigator — UCL St.Luc Brussels
Locations (2):
- Adult/Pediatric Limb Lengthening and Reconstruction - International Center for Limb Lengthening - Rubin Institute for Advanced Orthopedics Baltimore, Baltimore, Maryland, United States
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paley D. Congenital pseudarthrosis of the tibia: biological and biomechanical considerations to achieve union and prevent refracture. J Child Orthop. 2019 Apr 1;13(2):120-133. doi: 10.1302/1863-2548.13.180147. PMID 30996736
- [Background] Dufrane D. Impact of Age on Human Adipose Stem Cells for Bone Tissue Engineering. Cell Transplant. 2017 Sep;26(9):1496-1504. doi: 10.1177/0963689717721203. PMID 29113460